CLINICAL TRIAL: NCT02478957
Title: Randomized, Double-blind, Placebo-controlled, Crossover Design, Efficacy and Safety Study With PA101 in Patients With Indolent Systemic Mastocytosis
Brief Title: Treatment of Indolent Systemic Mastocytosis With PA101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patara Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA101-SM-02
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Mastocytosis; Systemic Mastocytosis; Indolent Systemic Mastocytosis
Keywords: mastocytosis; cromolyn sodium
MeSH Terms: conditions — Mastocytosis; Mastocytosis, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PA101 (Experimental): PA101, 40 mg administered via inhalation three times daily for 6 weeks
  Interventions: Drug: PA101
- Placebo (Placebo Comparator): Placebo, administered via inhalation three times daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PA101 — 40 mg PA101 administered via inhalation three times daily for 6 weeks
  Arms: PA101
Drug: Placebo — matching placebo administered via inhalation three times daily for 6 weeks
  Arms: Placebo

SUMMARY:
This is a randomized, placebo- and active-controlled, 2-period crossover, 2 cohort study in adult patients with indolent systemic mastocytosis (ISM).

The purpose of the study is to determine the efficacy and safety profile of PA101 delivered via eFlow high efficiency nebulizer in patients with ISM who are symptomatic despite using standard treatments.

DETAILED DESCRIPTION:
The symptom scores for determining eligibility will be established during the 2-week Run-in Period using eDiary and the eligible patients will be randomly allocated in a 2:1 ratio to one of two treatment cohorts at the baseline visit.

In Cohort 1 (n=24), patients will receive inhaled 40 mg PA101 three times daily and inhaled placebo three times daily via eFlow for 6 weeks each in a double-blind, 2-period crossover fashion with a 4-week washout period between the treatment periods.

In Cohort 2 (n=12), patients will receive inhaled 40 mg PA101 three times daily via eFlow and oral cromolyn sodium 200 mg four times daily for 6 weeks each in an open label, 2-period crossover fashion with a 4-week washout period between the treatment periods.

Patients will be allowed to use the same daily doses of pre-randomization H1 and H2 antihistamines as well as the same daily doses of any other allowed medications during each treatment period.

Visits during each treatment period will occur at the baseline Visit, and at the end of Weeks 1, 2, 4, and 6.

Blood and urine samples will be collected to test for various biomarkers. In a subset of patients, additional clinical assessments of the skin will be performed and blood samples will be collected for pharmacokinetic assessments. Clinical safety assessments will be performed in all patients at the start and end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of indolent systemic mastocytosis (ISM) according to the WHO criteria and the consensus proposal (2001)
* Experiencing at least one predefined qualifying symptom in at least two organ systems within 3 months of Screening despite the use of H1 and/or H2 antihistamines and other anti-mediator therapy
* Experiencing symptoms with a severity score of at least 4 for at least 7 out of 14 days during the Run-in period with at least one predefined qualifying symptom each from at least two organ systems, despite the use of H1 and/or H2 antihistamines and/or other anti-mediator therapy
* Willing and able to use an eDiary device daily for the duration of the study
* Completed at least 5 eDiary reports during each of two consecutive weeks of the Run-in period
* Willing and able to provide written informed consent prior to any study procedures

Exclusion Criteria:

* Advanced systemic mastocytosis (i.e., aggressive systemic mastocytosis [ASM], mast cell leukemia [MCL], or systemic mastocytosis with an associated clonal hematologic non-mast cell lineage disease [SM-AHNMD] )
* Current or recent history of clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine, psychiatric, malignant, or other illnesses that could put the patient at risk or compromise the quality of the study data as determined by the Investigator
* Use of oral cromolyn sodium within 6 weeks of Screening
* History of systemic corticosteroid, immunosuppressive, or anti-IgE monoclonal antibody therapy (e.g., omalizumab) within 6 months of Screening
* History of anaphylaxis requiring systemic treatment (i.e., corticosteroid or epinephrine) within 12 months of Screening
* Upper or lower respiratory tract infection within 4 weeks of Screening
* History of malignancy within the last 5 years, except basal cell carcinoma or cervix carcinoma in situ
* Major surgery within 6 months of Screening
* Current or recent history (within 12 months) of excessive use or abuse of alcohol
* Current or recent history (within 12 months) of abusing legal drugs or use of illegal drugs or substances
* Pregnant or breastfeeding females, or if of child-bearing potential unwilling to practice acceptable means of birth control or abstinence during the study
* Participation in any other investigational drug study within 4 weeks of Screening
* History of hypersensitivity or intolerance to aerosol medications or cromolyn sodium

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Overall symptom score | 6 weeks
  Mastocytosis Activity of Symptoms (MAS Plus) questionnaire for daily symptom score using eDiary

SECONDARY OUTCOMES:
Disease specific quality of life (QoL) | 6 weeks
  Mastocytosis Impact Questionnaire (MIQ) for quality of life
Patient Global Impression of Change (PGIC) scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Siebenhaar, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (8):
- Hopital Necker - Enfants Malades, Paris, France
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Darmstadt, Darmstadt
  - University Medical Center Mainz, Mainz
  - Technical University München, Munich
- University of Salerno, Salerno, Italy
- University Medical Center of Groningen, Groningen, Netherlands
- Hospital Universitario de Fuenlabrada, Madrid, Spain